CLINICAL TRIAL: NCT03487198
Title: A Phase 3, Multicenter, Randomized, Double-blind, Placebo-controlled Trial Evaluating the Safety and Efficacy of Brexpiprazole as Adjunctive Therapy in the Treatment of Major Depressive Disorder
Brief Title: The Safety and Efficacy of Brexpiprazole as Adjunctive Therapy in the Treatment of Major Depressive Disorder
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: In consideration of the progress now and the expected enrollment in the next few years,the NDA will not be acquired before the patent went out.
Sponsor: Otsuka Beijing Research Institute (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 331-403-00023
Record Dates: First submitted 2018-03-23; First posted 2018-04-03 (Actual); Last update posted 2020-12-29 (Actual); Status verified 2019-05

CONDITIONS: Major Depressive Disorder
Keywords: Major Depressive Disorder; Brexpiprazole
MeSH Terms: conditions — Depressive Disorder, Major | interventions — brexpiprazole

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Brexpiprazole (Experimental): 2-3 mg/day, once daily for 6 weeks, oral administration
  Interventions: Drug: Brexpiprazole
- Placebo (Placebo Comparator): 2-3 mg/day, once daily for 6 weeks, oral administration
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Brexpiprazole — Brexpiprazole 2-3mg/day
  Arms: Brexpiprazole
Drug: Placebo — Placebo 2-3 mg/day
  Arms: Placebo

SUMMARY:
This study is a multicenter, randomized, double-blind, placebo-controlled trial designed to assess the efficacy and safety of brexpiprazole as adjunctive therapy in the treatment of Major Depressive Disorder. A total of approximately 1100 subjects will be enrolled into the single-blind treatment for 6 weeks, and 480 incomplete responders will be randomized to brexpiprazole (2~3 mg) or placebo in a 1:1 ratio (approximately 240 subjects in each group), for treatment of 6 weeks.

DETAILED DESCRIPTION:
Screening phase: It can last up to 28 days and will begin when informed consent is signed. The screening phase will serve the following purposes: 1) To review the inclusion and exclusion criteria; 2) To allow for appropriate washout of prohibited medications; 3) To establish a pretreatment baseline of critical outcome measures.

Single-blind Prospective Treatment Phase (Phase A): It lasts 8 weeks; the purpose of the Phase A is to select the MDD subjects with incomplete response to ADT.

Randomized Double-blind Treatment Phase (Phase B): It lasts 6 weeks; the purpose of Phase B is to compare the efficacy and safety of Brexpiprazole as adjunctive therapy in the treatment of MDD patients with incomplete response to ADT.

Continued Treatment Phase after Phase A (Phase A+): It lasts 6 weeks; the purpose of Phase A+ is to continue treatment for subjects with complete response to ADT and not satisfying the criteria for Phase B.

Follow-up Phase: It lasts 4 weeks and only applies to the subjects from Phase B; the purpose of Follow-up Phase is to collect the safety information after the last dose of IMP.

ELIGIBILITY:
Inclusion Criteria:

1. The subject who are able to provide signed written informed consent.
2. Male and female outpatients 18 to 65 years of age, inclusive, at the time of signing the informed consent.
3. Subjects with both a diagnosis of MDD, and in a current Major Depressive Episode, according to the diagnostic criteria in DSM-IV-TR and confirmed by the Mini International Neuropsychiatric Interview (MINI). The current Major Depressive Episode must be ≥ 8 weeks in duration.
4. Subjects must have reported a history for the current Major Depressive Episode of an inadequate response to at least one and no more than three standard antidepressant treatments (including any antidepressants being received during Screening period, if the antidepressants treatment meets criteria of standard treatment). For the most recent antidepressant treatment, the subject must not report ≥ 50% improvement.

   Standard treatment is defined as: an antidepressant treatment for at least 6 weeks in duration (at least 3 weeks if combined treatment) at a minimum effective dose (or higher) according to prescription drug labels. At least once of 1 to 3 standard treatments is monotherapy for more than 6 weeks.

   An inadequate response is defined as: < 50% reduction in depressive symptom severity, as measured by the subject's self-report score on Visual Analogue Scale (VAS).
5. Subjects with a HAM-D17 Total Score ≥ 18 at the Screening and Baseline visits.

Phase B (Double-blind Randomization Phase)

At the end of Phase A (Week 8 visit), the subjects entering Phase B should also meet all of the following inclusion criteria (criteria for incomplete response):

1. HAM-D17 total score ≥14 at the end of phase A.
2. < 50% reduction in HAM-D17 total score at the end of phase A (end of Week 8) relative to baseline.
3. A CGI-I score ≥ 3 at Weeks 2, 4, 6, and 8.

Exclusion Criteria:

1. Females of childbearing potential and male subjects who are not willing to or cannot practice contraceptive methods during the trial and for 30 days after the last dose.
2. Females who are breast-feeding or lactating and who have a positive pregnancy test result (Urine or serum test) prior to screening or randomization (within 72 hours).
3. Subjects who report treatment with adjunctive antipsychotic medication with an antidepressant during the current Major Depressive Episode.
4. Subjects who report allergies or an intolerability to all protocol-specified ADTs or subjects with contraindication for protocol-specified ADTs described in their prescription drug labels.
5. Subjects who have had an ECT treatment history at any time in the past or at present, or who have had a vagus nerve stimulation or deep brain stimulation device implanted for management of treatment-resistant depression.
6. Subjects with a current need for hospitalization or who have been hospitalized within four weeks prior to screening for the current Major Depressive Episode.
7. Subjects with a current Axis I (DSM-IV-TR) diagnosis of:

   * Delirium, dementia, amnestic or other cognitive disorder
   * Schizophrenia, schizoaffective disorder, or other psychotic disorder
   * Bipolar I or II disorder
   * Eating disorder (including anorexia nervosa or bulimia)
   * Obsessive compulsive disorder
   * Panic disorder
   * Post-traumatic stress disorder
8. Subjects with a current Axis II (DSM-IV-TR) diagnosis of borderline, antisocial, paranoid, schizoid, schizotypal or histrionic personality disorder.
9. Subjects experiencing hallucinations, delusions or any psychotic symptomatology in the current Major Depressive Episode.
10. Subjects who have met DSM-IV-TR criteria for substance abuse or dependence within the past 180 days prior to screening; including alcohol and benzodiazepines, but excluding caffeine and nicotine.
11. Subjects receiving new onset psychotherapy (individual, group, marriage, or family therapy) within 6 weeks of screening or at any time during participation in the trial.
12. Subjects who present a serious risk of suicide.

    * Subjects who answer "Yes" on the C-SSRS Suicidal Ideation Item 4 and whose most recent episode meeting criteria for this C-SSRS Item 4 occurred within the last 6 months; OR
    * Subjects who answer "Yes" on the C-SSRS Suicidal Ideation Item 5 and whose most recent episode meeting criteria for this C-SSRS Item 5 occurred within the last 6 months; OR
    * Subjects who answer "Yes" on any of the 5 C-SSRS Suicidal Behavior Items (actual attempt, interrupted attempt, aborted attempt, preparatory acts or behaviors, or suicidal behavior) and whose most recent episode meeting criteria for any of these 5 C-SSRS Suicidal Behavior Items occurred within the last 2 years; OR
    * Subjects who, in the opinion of the investigator, present a serious risk of suicide.
13. Medical history or clinical evidence (abnormal clinical significant laboratory test, vital signs, or ECG findings, judged by investigator) shows the health condition of the subject may cause an undue adverse event or interfere with assessments of safety/efficacy during the course of the trial.
14. Subjects with a history of ischemic heart disease or myocardial infarction, congestive heart failure (whether controlled or uncontrolled), angioplasty, stenting, or coronary artery bypass surgery.
15. Subjects with insulin-dependent diabetes mellitus (IDDM, i.e., any subjects using insulin) and uncontrolled non-IDDM are excluded. Subjects with non-IDDM may be eligible for the trial if their condition is stable as determined by satisfying ALL of the following criteria:

    * Glycosylated hemoglobin (HbA1c) < 7.0%, AND
    * Screening glucose must be ≤ 125 mg/dL or ≤ 6.94 mmol/L (fasting) or <200 mg/dL or <11.1 mmol/L (non-fasting). If the non-fasting screening glucose is ≥ 200 mg/dL or ≥ 11.1 mmol/L, subjects must be retested in a fasted state and the retest value must be ≤ 125 mg/dL or ≤ 6.94 mmol/L, AND
    * Subject has been maintained on a stable regimen of oral anti-diabetic medication(s) for at least 28 days prior to screening or diabetes has been well-controlled by diet for at least 28 days prior to screening, AND
    * Subject has not had any hospitalizations within the 12 months prior to screening due to diabetes or complications related to diabetes, AND
    * Subject's diabetes is not newly diagnosed during screening for the trial.
16. Subjects with hypothyroidism or hyperthyroidism (unless condition has been stabilized with medications for at least the past 90 days) and/or an abnormal result for free T4 at screening. Eligibility of subjects excluded based on an abnormal free T4 result can be discussed with the medical monitor if, in the investigator's judgment, the subject is a suitable candidate for the trial.
17. Subjects with a history of neuroleptic malignant syndrome (NMS) or 5-HT syndrome.
18. Subjects with a history of true allergic response (i.e., not intolerance) to more than one class of medications.
19. Subjects with epilepsy or a history of seizures, except for a single seizure episode, for instance childhood febrile seizure, post traumatic, or alcohol withdrawal.
20. Subjects with uncontrolled hypertension (diastolic blood pressure [DBP] > 95 mmHg in any position) or symptomatic hypotension, or orthostatic hypotension which is defined as a decrease of ≥ 30 mmHg in systolic blood pressure (SBP) and/or a decrease of ≥ 20 mmHg in DBP after at least 3 minutes standing compared to the previous supine blood pressure, OR development of symptoms.
21. The following laboratory test and ECG results are exclusionary:

    * QTc ≥ 450 msec (for males) or ≥ 470 msec (for females) in ECG
    * Platelets ≤75×109/L (7,5000/mm3)
    * Hemoglobin ≤90 g/L (9 g/dL)
    * Neutrophils ≤1×109/L (1,000/ mm3)
    * AST or ALT > 2 ×upper limit of normal (ULN)
    * Creatinine ≥ 2 mg/dL
    * Creatine phosphokinase (CPK) > 3 × ULN
    * HbA1c ≥ 7.0%
22. Treatment with MAOI (e.g., Nardil® [phenelzine]) within the 2 weeks prior to the start of Phase A.
23. Use of benzodiazepines and/or hypnotics (including non-benzodiazepine sleep aids) within 1 week prior to the start of Phase A, but excluding short-acting non-benzodiazepine sleep aids (ie, zolpidem, zaleplon, zopiclone, and eszopiclone only).
24. Subjects who participated in a clinical trial within the past 90 days or who participated in more than two clinical trials within the past year.
25. Any subject who, in the opinion of the investigator, should not participate in the trial. Such as, any subject who is impossible to compliance with the protocol, or who would be likely to require prohibited concomitant medication/therapy during the trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2018-05-30 (Actual); Primary Completion 2019-05-30 (Actual); Study Completion 2019-05-30 (Actual)

PRIMARY OUTCOMES:
Change from the end of Phase A (Week 8 visit) to the end of Phase B (Week 14 visit) in the MADRS Total Score | Week 8 and Week 14
  The objective of the primary analysis is to compare the efficacy of brexpiprazole (2~3 mg/day) to placebo as adjunctive therapy to an assigned open-label ADT in adult subjects with MDD who demonstrate an incomplete response after 8 weeks of treatment with the same assigned open-label antidepressant therapy (ADT). The efficacy is assessed by the change from the end of Phase A (Week 8 visit) to the end of Phase B (Week 14 visit) in the MADRS Total Score

SECONDARY OUTCOMES:
Change from the end of Phase A (Week 8 visit) to the end of Phase B (Week 14 visit) in SDS Mean Score | Week 8 and Week 14
  The efficacy is assessed by the change from the end of Phase A (Week 8 visit) to the end of Phase B (Week 14 visit) in SDS Mean Score
Change from the end of Phase A (Week 8 visit) in MADRS Total Score for every trial week visit in Phase B other than Week 14 visit | Week 8 and Week 14
  The efficacy is assessed by the change from the end of Phase A (Week 8 visit) in MADRS Total Score for every trial week visit in Phase B other than Week 14 visit
Change from the end of Phase A (Week 8 visit) for every trial week visit in Phase B in CGI - Severity of Illness scale (CGI-S) score | Week 8 and Week 14
  The efficacy is assessed by the Change from the end of Phase A (Week 8 visit) for every trial week visit in Phase B in CGI - Severity of Illness scale (CGI-S) score
Change from the end of Phase A (Week 8 visit) to the end of Phase B (Week 14 visit) in HAM-D17 Score | Week 8 and Week 14
  The efficacy is assessed by the change from the end of Phase A (Week 8 visit) to the end of Phase B (Week 14 visit) in HAM-D17 Score
CGI - Improvement scale (CGI-I) score for every trial week visit in Phase B | Week 8 and Week 14
  The efficacy is assessed by the CGI-I score for every trial week visit in Phase B
MADRS Response Rate at every trial week visit in Phase B | Week 8 and Week 14
  The efficacy is assessed by the MADRS Response Rate at every trial week visit in Phase B, where response is defined as ≥ 50% reduction in MADRS Total Score from the end of Phase A (Week 8 visit)
CGI-I Response rate at every trial week visit in Phase B | Week 8 and Week 14
  The efficacy is assessed by the CGI-I Response rate at every trial week visit in Phase B, where response is defined as a CGI-I score of 1 or 2 (very much improved or much improved)
Change from the end of Phase A (Week 8 visit) to the end of Phase B (Week 14 visit) in 16-item Quick Inventory of Depressive Symptomatology Self-Report (QIDS-SR16) Score | Week 8 and Week 14
  The efficacy is assessed by the Change from the end of Phase A (Week 8 visit) to the end of Phase B (Week 14 visit) in QIDS-SR16 Score
QIDS-SR16 Response Rate at every trial week visit in Phase B | Week 8 and Week 14
  The efficacy is assessed by the QIDS-SR16 Response Rate at every trial week visit in Phase B, where response is defined as ≥ 50% reduction in QIDS-SR16 Total Score from the end of Phase A (Week 8 visit)
QIDS-SR16 Complete Remission Rate (recovery) at every trial week visit in Phase B | Week 8 and Week 14
  The efficacy is assessed by the QIDS-SR16 Complete Remission Rate (recovery) at every trial week visit in Phase B, where complete remission (recovery) is defined as QIDS-SR16 Total Score ≤ 5

CONTACTS AND LOCATIONS:
Overall Officials: Patyman Juma, Study Director — Otsuka Beijing Research Institute
Locations (1):
- Beijing Anding Hospital of Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No